CLINICAL TRIAL: NCT07339410
Title: Effects of Manual Therapy and Structured Exercises on Postural Balance and Walking Capacity in Adults With Hemophilia
Brief Title: Physiotherapy to Improve Balance and Walking Capacity in Hemophilia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Ayse Merve TAT, Assistant Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YuzuncuYil2026
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Hemophilia
Keywords: Manual therapy; Exercise; Postural balance; walking; hemophilia; arthropathy
MeSH Terms: conditions — Hemophilia A; Motor Activity; Joint Diseases | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention)
- Physiotherapy Group (Experimental): Physiotherapy
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — The physiotherapy intervention applied in this study included manual therapy and a structured and progressive exercise program.
  Arms: Physiotherapy Group

SUMMARY:
Introduction: Hemarthrosis is the most common type of bleeding with 70-80% in patient with hemophilia (PwH) and the majority of hemarthrosis occurs in the knee and ankle joints. Recurrent hemarthrosis may cause pain, limited range of motion (ROM), atrophy, swelling, crepitus, and decreased proprioceptive sensation and ultimately causes hemophilic arthropathy. Preventing hemarthrosis and treating arthropathy symptoms in PwH may improve static and dynamic balance and walking capacity. The aim of this study was to investigate the effects of manual therapy and structured exercises on joint health, activity pain, walking capacity and static and dynamic balance.

Method: Thirty-five AwH were randomly assigned to two groups using the computerised simple randomization method: the control group (CG) and the physiotherapy group (PG). The sample sizes for the CG and PG are 17 and 18, respectively. Hemophilia type and severity, treatment regime (prophylaxis or on-demand), age, height and weight were recorded. Joint health was assessed with Hemophilia Joint Health Score (HJHS) version 2.1 by a hemophilia specialist physiotherapist. Activity pain was assessed with Numeric Pain Scale (NPS). Walking capacity was evaluated 6 Minute Walking Test (6MWT). Postural balance (static and dynamic balance) were evaluated with the Pro-kin Technobody Posturographic Platform (Pro-kin 212, Technobody s.r.l, Dalmine, 21044 Bergamo, Italy). Static stability test was used for static balance assessment. Dynamic balance was evaluated with the Limits of Stability (LoS) test. The PG received 12 physiotherapy sessions twice a week for 6 weeks. The physiotherapy intervention consisted of manual therapy and a structured, progressive exercise program. The CG continued with their routine hemophilia care.

ELIGIBILITY:
Inclusion Criteria:

* Severe or moderate hemophilia A or B
* Aged 18-65
* Having at least 3 points from at least one of the knee and ankle index joints in the Hemophilia Joint Health Score
* Volunteering to attend physiotherapy sessions regularly

Exclusion Criteria:

* Receiving physiotherapy or undergone surgery on lower extremity within the last 6 months
* Having neurological or cognitive disease
* Having visual and vestibular system pathologies

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2025-10-20 (Actual); Primary Completion 2025-12-20 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Postural balance | From enrollment to the end of treatment at 6 weeks
  Static and dynamic postural balance were evaluated with the Pro-kin Technobody Posturographic Platform (Pro-kin 212, Technobody s.r.l, Dalmine, 21044 Bergamo, Italy).
Walking capacity | From enrollment to the end of treatment at 6 weeks
  Walking capacity was evaluated with 6 Minute Walking Test.

SECONDARY OUTCOMES:
Activity pain | From enrollment to the end of treatment at 6 weeks
  Activity pain was evaluated with Numeric Pain Scale
Joint health | From enrollment to the end of treatment at 6 weeks
  Joint health was evaluated with Hemophilia Joint Health Score

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yüzüncü Yıl University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided